CLINICAL TRIAL: NCT01312363
Title: A Six-month, Open Labeled, Multi-centered, Observational Study for the Tolerability of Exelon Patch (Rivastigmine) for Patients With Alzheimer's Disease
Brief Title: Study for the Tolerability of Exelon Patch (Rivastigmine) for Alzheimer's Disease (AD) Patients
Acronym: X-MEN
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul St. Mary's Hospital (Other); Korea University (Other); Bobath Memorial Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Hanyang University (Other); Kwandong University Myongji Hospital (Unknown); Inha University Hospital (Other); SungAe General Hospital (Unknown); Ewha Womans University (Other); Inje University (Other); Hanyang University Seoul Hospital (Other); Kyunghee University Medical Center (Other); Hallym University Medical Center (Other); Pusan National University Hospital (Other); Konyang University Hospital (Other); Wonkwang University Sanbon Medical Center (Unknown); Yong-in Hyoja Geriatric Hospital (Unknown); Jeju National University (Other); Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, SangYun Kim, Department of Neurology, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seoul National University Hospital
Other Study IDs: X-MEN
Record Dates: First submitted 2010-10-26; First posted 2011-03-10 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Rivastigmine; Patch; Tolerability
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rivastigmine patch — Rivastigmine patch (5-10cm2, daily, 24hr)
  Other Names: Exelon patch

SUMMARY:
The investigators plan to see what factors can influence the durability of Exelon patch treatment in Korean patients with Alzheimer's disease.

Based on these results, the investigators will find the ways to maximize the effect and durability of Exelon patch on Korean patients with Alzheimer's disease.

After finishing this study, the investigators are going to present the study results at the international and national academic meetings or conferences.

Also the investigators expect that they can publish the result in a journal of in the field of neurology or dementia till the winter of 2010.

DETAILED DESCRIPTION:
A once-daily Exelon patch has recently been developed to reduce the GI side effect of rivastigmine and make application easier by once a day.

Thinking the patch as the first-line drug, it should be proven as safe for a long time. The safety and clinical effect of Exelon patch was tested in many studies.

However, most of studies have been conducted on Western countries and the study period was not more than a year.

There are only few data on Exelon patch related to other ethnic such as Asian patients with Alzheimer's disease.

Especially, there are many different environmental factors between Western and Asia countries, such as habitual or climate factors, skin type and behavioral styles which may be influenced on patch durability.

The aim of this study was to evaluate the durability of Exelon patch in Korean patients with Alzheimer's disease and what are the factors influencing the durability.

Also evaluating the significance of factors gives us the way to increase the patch durability.

Thirty patients per investigational center will be enrolled during 6 months.

Probable mild to moderate AD patients will be included whether they have depression or other neurological symptoms or diseases.

The period of this study will be 6 months, and we will start the treatment starting from Exelon patch 5cm2.

After 4 weeks, dose titration will be attempted to Exelon patch 10cm2.

If a patient is reporting too much discomfort to stick on high dose patch, investigators will assess the severity of the side effects followed by adjusting dose or considering discontinuation.

Cognitive, functional, and global outcome measures are obtained at baseline and at the end of month 6. Environmental factors including caregiver condition, participant's habitat type, and participant's skin type, etc. are also evaluated from the first visit, and they will be assessed at every visit.

Participants and their caregivers will be asked of any possible concerns or problems associated with patch use at every visit. And if there is any visible problem or adverse event, it will be taken as a picture and be uploaded to investigation web site for this study.

Finally, for the primary endpoint, participants who discontinue prematurely are evaluated during every visit.

Signs of skin irritation at the site of patch application are assessed at every visit by the investigator using skin irritation rating scale.

Caregivers evaluate patch adhesion throughout the study with ratings provided in accordance with a patch adhesion scoring system.

To assess factors to influence skin irritation or any other adverse events, we will classify skin type of each participant using "skin type measuring paper" at the first visit time.

We will search for any personal or family history of allergy, and characteristics of participant's habitat using questionnaire.

The information about the caregiver including his/her condition based on the annual income, living status, and education level.

To see if there is any specific allergic factor for discontinuation, we will investigate participant's allergy history more completely and thoroughly.

ELIGIBILITY:
Inclusion Criteria:

* Probable AD by NINCDS-ADRDA and DSM-IV
* Male and female aged from 51 to 85 years old
* Magnetic resonance imaging or computed tomographic scan within 12 months consistent with a diagnosis of probable AD
* Patients who approved to release of personal information

Exclusion Criteria:

* Patient with any active pulmonary, gastrointestinal, renal, hepatic (severe hepatic function impaired patients), endocrine, or cardiovascular disease, clinically significant laboratory abnormalities, or any medical condition which would prohibit them from completing the study
* Any patients suspicious of drug addiction or alcohol addiction for the past 10 years
* Any other patients to be decided to be inappropriate for the study by the investigators

Ages: 51 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 24 weeks
  number of participants with skin irritation or other adverse events

SECONDARY OUTCOMES:
Factors for the disuse of Rivastigmine patch | 24 weeks
  to search for the factors that affect the disuse of Rivastigmine patch in each patient, such as skin irritation,abnormal clinical laboratory factors, or environmental factors.

CONTACTS AND LOCATIONS:
Overall Officials: SangYun Kim, MD, PhD, Study Chair — Seoul National University College of Medicine & Seoul National University Bundang Hospital; Dong Won Yang, MD, PhD, Study Director — The Catholic University of Korea; Moon Ho Park, MD, PhD, Study Director — Korea University College of Medicine & Korea University Ansan Hospital; Hae Ri Na, MD, Study Director — Bobath Memorial Hospital; Young-Chul Yoon, MD, PhD, Principal Investigator — Chungang University College of Medicine & Chungang University Hospital; Seong-Ho Koh, MD, PhD, Principal Investigator — Hanyang University College of Medicine & Hanyang University Guri Hospital; Hyun Jeong Han, MD, PhD, Principal Investigator — Kwandong University College of Medicine & Myongji Hospital; Bon D. Ku, MD, PhD, Principal Investigator — Kwandong University College of Medicine & Myongji Hospital; Seong-Hye Choi, MD, PhD, Principal Investigator — Inha University College of Medicine & Inha University Hospital; Jung Seok Lee, MD, Principal Investigator — Jeju National University College of Medicine & Jeju National University Hospital; Jun-Seong Lim, MD, Principal Investigator — SungAe General Hospital; Jung Eun Kim, MD, Principal Investigator — Ewha Womans University School of Medicine & Ewha Womans University Mokdong Hospital; Jeong Yeon Kim, MD, Principal Investigator — Inje University College of Medicine & Sanggye Paik Hospital; Hee-Jin Kim, MD, Principal Investigator — Hanyang University College of Medicine & Hanyang University Seoul Hospital; Seung Hyun Kim, MD, PhD, Principal Investigator — Hanyang University College of Medicine & Hanyang University Seoul Hospital; Key Hung Park, MD, PhD, Principal Investigator — Kyung Hee University College of Medicine & Kyung Hee University Medical Center; Kyung Won Park, MD, PhD, Principal Investigator — Dong-A University College of Medicine & Dong-A University Medical Center; Hui Chul Choi, MD, PhD, Principal Investigator — Hallym University College of Medicine & Hallym University Chunchon Hospital; Eun-Joo Kim, MD, Principal Investigator — Pusan National University School of Medicine & Pusan National University Hospital; Bora Yoon, MD, Principal Investigator — Konyang University School of Medicine & Konyang University Hospital; Hyun Duk Yang, MD, Principal Investigator — Wonkwang University College of Medicine & Wonkwang University Sanbon Medical Center; Youngsoon Yang, MD, Principal Investigator — Yong-in Hyoja Geriatric Hospital; Hee-Jung Seo, MD, Principal Investigator — Yong-in Hyoja Geriatric Hospital
Locations (19):
- South Korea (19):
  - Dong-A University Hospital, Busan, Busan
  - Pusan National University Hospital, Busan, Busan
  - Hallym University Chunchon Hospital, Chunchon, Chunchon
  - Konyang University Hospital, Daejeon, Daejeon
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Wonkwang University Sanbon Medical Center, Gunpo, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Bobath Memorial Hospital, Seongnam-si, Gyeonggi-do
  - Yong-in Hyoja Geriatric Hospital, Yongin-si, Gyeonggi-do
  - Inha University Hospital, Incheon, Incheon
  - Jeju National University Hospital, Jeju City, Jeju-do
  - Seoul St. Mary's Hospital, Seoul, Seoul
  - SungAe General Hospital, Seoul, Seoul
  - Chungang University Hospital, Seoul, Seoul
  - Ewha Womans University Hospital, Seoul, Seoul
  - Hanyang University Seoul Hospital, Seoul, Seoul
  - Kyung Hee University Medical Center, Seoul, Seoul
  - Sanggye Paik Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: Undecided